CLINICAL TRIAL: NCT07328087
Title: COLONYVAQ™-CRC, a Physics-aware, Quantum-Classical AI-Guided Personalized Neoantigen Peptide Vaccine, Administered in Combination With Standard Adjuvant Oxaliplatin-based Chemotherapy (mFOLFOX6 or CAPOX) and Nivolumab 3 mg/kg in Patients With Completely Resected Stage III Microsatellite-stable (MSS)
Brief Title: COLONYVAQ™, a Quantum-Classical Guided Personalized Neoantigen Vaccine for MSS Stage III Colorectal Cancer
Acronym: COLONYVAQ™-CRC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Biogenea Pharmaceuticals Ltd. (Industry)
Collaborators: Interbalkan Medical Center, Thessaloniki, Greece (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BiogeneaTMMyVaccine3; 10210381179 (Other Grant/Funding Number: Biogenea™ Pharmaceuticals Ltd); COLONYVAQ-CRC P1-Adjuvant-MSS™ (Other: Myoncotherapy™)
Record Dates: First submitted 2025-12-05; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Metastatic; Colorectal Cancer Stage III; Colorectal Cancer Stage IV
Keywords: CRC Patient-specific vaccine,; AI-Quantum guided neoantigen selection,; Machine learning-based neoantigen prediction,
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Twelve patients will enroll in the initial safety cohort. If, among these 12 patients, fewer than 3 experience toxicity greater than grade II (grade III or IV) attributed to the experimental vaccine preparation and no patient experiences experimental-preparation-related grade IV toxicity, the study will expand to enroll a total of 50 patients. If these criteria are not met, the protocol and dose/schedule may be revised and further enrollment paused or modified.
  Estimated Enrollment: 12 patients in the initial safety phase; up to 50 patients in total upon expansion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm: COLONYVAQ-CRC + Standard Adjuvant Chemotherapy + Nivolumab (Experimental): All enrolled patients receive study treatment after R0 resection of stage III MSS/pMMR colorectal cancer. Standard adjuvant chemotherapy is either mFOLFOX6 or CAPOX, preselected per institutional practice. mFOLFOX6 is given q14d for ~6 months: oxaliplatin 85 mg/m² IV over 2 h, leucovorin 400 mg/m² IV over 2 h, 5-FU 400 mg/m² IV bolus, then 5-FU 2400 mg/m² continuous IV over 46 h. CAPOX is given q21d for ~3-6 months: oxaliplatin 130 mg/m² IV over ~2 h on Day 1 plus capecitabine 1000 mg/m² PO BID on Days 1-14, then 7 days off. COLONYVAQ-CRC is a personalized multi-peptide neoantigen vaccine (≤20 peptides, 8-30 aa, 0.3 mg each), selected by a quantum-classical pipeline, synthesized under GMP, pooled (2-4 pools) and mixed 1:1 with poly I:C (2 mg/mL) to 1 mL for SC injection on a prime-boost schedule (Days 1, 4, 8, 15, 22; Weeks 12, 20). Nivolumab 3 mg/kg IV q2w is given for up to 12 months.
  Interventions: Biological: Experimental: COLONYVAQ-CRC + mFOLFOX6 or CAPOX + Nivolumab

INTERVENTIONS:
Biological: Experimental: COLONYVAQ-CRC + mFOLFOX6 or CAPOX + Nivolumab — Intervention Type: Biological Intervention Name: COLONYVAQ-CRC (Personalized Neoantigen Peptide Vaccine)
  Description:
  COLONYVAQ-CRC is a personalized multi-peptide neoantigen vaccine composed of up to 20 patient-specific synthetic peptides (8-30 amino acids; 0.3 mg per peptide per dose). Neoantigens are selected from tumor/normal whole-exome and tumor RNA sequencing using the COLONYVAQ quantum-classical pipeline (including HLA typing, quantum-geometric similarity, thermodynamic docking, and calibrated immunogenicity scoring). Peptides passing all physics-immunology gates are synthesized under GMP, grouped into 2-4 pools (≤5 peptides/pool in 500 µL), and mixed 1:1 with Montamide (2 mg/mL) to a final volume of 1 mL for subcutaneous injection into lymph node-rich regions (e.g., bilateral axillae/groins). Vaccination follows a prime-boost schedule (e.g., Days 1, 4, 8, 15, 22; booster doses around Weeks 12 and 20), coordinated with chemotherapy.

SUMMARY:
This is an early phase I, single-arm, open-label clinical study designed to evaluate the safety, tolerability, and feasibility of COLONYVAQ-CRC, a physics-aware, quantum-classical AI-guided personalized neoantigen peptide vaccine, administered in combination with standard adjuvant oxaliplatin-based chemotherapy (mFOLFOX6 or CAPOX) and nivolumab 3 mg/kg in patients with completely resected stage III microsatellite-stable (MSS) / proficient mismatch repair (pMMR) colorectal cancer. An initial safety cohort of 12 patients will be enrolled and closely monitored for toxicity attributable to the experimental vaccine preparation. If, among these 12 patients, fewer than 3 develop experimental-preparation-related toxicity greater than grade 2 and no patient develops experimental-preparation-related grade 4 toxicity, the study will expand to enroll a total of 50 patients. Primary objectives focus on safety and tolerability of the combination regimen. Secondary and exploratory objectives characterize neoantigen-specific immune responses, ctDNA dynamics, T-cell receptor (TCR) clonotype evolution, tumor immune microenvironment features, and preliminary disease control (disease-free survival and overall survival) to inform subsequent phase II design.

DETAILED DESCRIPTION:
Colorectal cancer is a leading cause of cancer-related mortality. In stage III disease, recurrence remains frequent despite curative-intent surgery and adjuvant oxaliplatin-based chemotherapy. Immune checkpoint inhibitors have transformed outcomes in mismatch repair-deficient / microsatellite instability-high colorectal cancer, but microsatellite-stable / pMMR tumors typically exhibit a lower tumor mutational burden and a poorly inflamed, immunosuppressive microenvironment. As a result, conventional PD-1 blockade alone provides minimal benefit in MSS/pMMR disease. Earlier vaccine approaches in colorectal cancer focused on tumor-associated antigens such as CEA, MUC1, survivin, MAGE and multi-TAA peptide cocktails. These studies showed that peptide and dendritic-cell-based vaccines can induce antigen-specific T-cell and B-cell responses, yet objective responses were rare, clinical benefit was modest, and off-tumor toxicities were a concern because TAAs are frequently expressed in normal tissues. Tumor-specific neoantigens, generated by non-synonymous somatic mutations, are in contrast restricted to malignant cells, escape central tolerance, can elicit higher-avidity T-cell responses, and minimize off-tumor toxicity. Early colorectal and pan-cancer neoantigen trials, as well as shared-neoantigen programs such as SLATE-KRAS and fully personalized viral-RNA platforms such as GRANITE, have demonstrated that multi-neoantigen vaccination is feasible, safe, and immunogenic, particularly in low-burden or maintenance settings and when combined with checkpoint blockade. The adjuvant neoantigen dendritic cell vaccine plus nivolumab trial in resected hepatocellular carcinoma and colorectal liver metastases further supports the idea that personalized neoantigen vaccination in the minimal residual disease (MRD) setting can augment neoantigen-specific T-cell responses and potentially improve relapse-free survival. Oxaliplatin-based regimens (mFOLFOX6 or CAPOX) can induce immunogenic cell death, exposing calreticulin and other danger signals that enhance dendritic cell uptake and cross-presentation of tumor antigens. Nivolumab, by blocking PD-1, relieves inhibitory signaling on activated T cells. Combining a personalized multi-neoantigen peptide vaccine with immunogenic chemotherapy and PD-1 blockade is therefore expected to increase antigen release, improve antigen presentation, and augment effector function, potentially converting immunologically "cold" MSS tumors into more inflamed, "hot" lesions amenable to durable immune surveillance in the adjuvant setting.

COLONYVAQ-CRC: Quantum-Classical, Physics-Aware Neoantigen Prioritization Most existing neoantigen pipelines treat epitope ranking as mainly statistical. COLONYVAQ-CRC introduces a physics-aware, quantum-classical AI layer, adapted from Tamavaq, to generate an auditable, mechanistic chain from sequencing to clinical peptide selection. For each candidate peptide-HLA pair p, the system constructs a unified feature representation Φ(p), which concatenates sequence-based, biological, quantum, structural, and energetic evidence: Φ(p)=[e_"CNN" (p),"" aux(p),"" z_Q (p),"" ϕ_"struct" (p),""ϕ_"dock" (p)]. The term e_"CNN" (p) denotes a deep sequence/HLA embedding derived from convolutional or transformer models trained on large immunopeptidome datasets. The auxiliary block aux(p) compiles antigen processing and expression priors such as proteasomal cleavage likelihood, TAP transport propensity, transcript abundance, clonality and, when available, ctDNA/MRD information to approximate the effective antigen source strength. The quantum descriptor z_Q (p) is a low-dimensional classical vector that parameterizes a quantum circuit embedding. The structural term ϕ_"struct" (p) summarizes pocket occupancy and residue-residue contacts in modeled peptide-HLA complexes. Finally, ϕ_"dock" (p) aggregates docking ensemble statistics including pose energies, dispersion and conformational diversity.

Similarity between two candidates p and q is captured by a composite positive semi-definite kernel K_"total" (p,q)=αK_"CNN" (p,q)+βK_"aux" (p,q)+γK_Q (p,q)+δK_"struct" (p,q)+εK_"dock" (p,q), where the non-negative weights α,β,γ,δ,ε adjust the relative contribution of each modality. Because each component kernel is constructed to be positive semi-definite, their non-negative linear combination remains positive semi-definite, ensuring that K_"total" can be used consistently in kernel logistic regression or related methods. A decision function can be written as f(p)=∑_(i=1)^M▒α_i K_"total" (p,p_i)+b, where {p_i } are training peptides and α_i,b are learned coefficients. The immunogenicity probability is then modeled as I ̂(p)=σ(f(p)), where σ(z)=1/(1+e^(-z)) is the logistic function. On the quantum side, each peptide x is encoded as a normalized state ∣ψ(x)⟩ in a Hilbert space H of dimension 2^n, constructed via a feature map U(z_Q (x),θ) acting on a reference state ∣0⟩^(⊗n): ∣ψ(x)⟩=U(z_Q (x),θ)" "∣0⟩^(⊗n). The overlap between two peptide states is ⟨ψ(x)∣ψ(y)⟩. Quantum-geometric similarity is quantified by the Fubini-Study distance d_"FS" (x,y)=arccos⁡(∣⟨ψ(x)∣ψ(y)⟩∣), which lies in [0ⓜ,π/2], where d_"FS" =0 corresponds to identical rays and d_"FS" =π/2 to orthogonal states. From this distance, a quantum similarity kernel is defined as K_q (x,y)=〖∣⟨ψ(x)∣ψ(y)⟩∣〗^2=〖cos⁡〗^2 (d_"FS" (x,y)). This kernel can be interpreted as the probability that the state ∣ψ(x)⟩ is projected onto ∣ψ(y)⟩. When low-sequence-identity peptides share higher-order physicochemical structure, they may map to nearby points on this complex projective manifold, generating large K_q values even when classical sequence similarity is low. The internal structure and entanglement of ∣ψ(x)⟩ are monitored by forming reduced density matrices on subsystems. For a bipartition into subsystems A and B, the reduced state is ρ_A (x)=Tr_B (∣ψ(x)⟩⟨ψ(x)∣). The von Neumann entropy S_A (x)=-Tr[ρ_A (x)log⁡ρ_A (x)] quantifies entanglement between A and B. A regularization term encourages entropy within a target range, avoiding trivial product states (too little entanglement) and excessively entangled states that can be numerically unstable and difficult to approximate on noisy intermediate-scale quantum (NISQ) hardware.

The sensitivity of the quantum embedding to parameter changes is characterized by the quantum Fisher information matrix F(θ) with entries F_ij (θ)=R[⟨∂_i ψ∣∂_j ψ⟩-⟨∂_i ψ∣ψ⟩⟨ψ∣∂_j ψ⟩], where ∣∂_i ψ⟩=∂∣ψ(θ)⟩/∂θ_i. Ill-conditioned Fisher matrices, with very small eigenvalues, can lead to large variances in parameter estimates and unstable kernel values. COLONYVAQ therefore introduces a penalty proportional to tr(F(θ)^(-1)), which diverges when eigenvalues approach zero; minimizing this term nudges optimization toward parameter regions where all directions in parameter space are well informed by the data. Energetics are treated in a thermodynamically calibrated way. For each peptide-HLA docking pose i with standard free energy ΔG_i^∘, the microstate association and dissociation constants are K_(a,i)=exp⁡(ⓜ (ΔG_i^∘)/RT),K_(d,i)=exp⁡((ΔG_i^∘)/RT), with R=1.987×10^(-3) " " kcal⋅mol^(-1)⋅K^(-1) and T=310"" K, such that RT≈0.616" " kcal⋅mol^(-1). The docking ensemble is summarized as a Boltzmann-weighted effective association constant K_a^"eff" =∑_i▒w_i exp⁡(ⓜ-(ΔG_i^∘)/RT),∑_i▒w_i =1, yielding an effective free energy ΔG_"eff" ^∘=-RTln⁡K_a^"eff" and corresponding dissociation constant K_d^"eff" =1/K_a^"eff" . These values are reported in units familiar to experimentalists (kcal·mol-¹ for ΔG_"eff" ^∘, nM for K_d^"eff" ). If the spread of free energies in the ensemble is σ_ΔG, then the associated uncertainty in K_dcan be expressed multiplicatively as exp⁡(±σ_ΔG/(RT)). For example, at T=310"" K, a change of 1.2"" kcal⋅mol^(-1) in ΔG^∘ changes K_d by a factor of approximately exp⁡(1.2/0.616)≈6.3. A docking loss term L_"dock" =λ_1 E ˉ+λ_2 σ_E, where E ˉ and σ_E are the mean and standard deviation of docking energies, biases the model toward low-energy, low-variance ensembles that are empirically associated with robust peptide-MHC display. On top of Φ(p) and the kernel K_"total" , COLONYVAQ trains a calibrated logistic head I ̂(p)=σ(w^⊤ Φ(p)+b), which is interpreted as the probability that peptide p is recognized by T cells, optimized for both discrimination (for example AUC) and calibration (for example Brier score, expected calibration error). In parallel, a linear thermodynamic head predicts (ΔG) ̂^∘ (p)=η^⊤ Φ(p)+η_0, from which a predicted dissociation constant K ̂_d (p)=exp⁡((ΔG) ̂^∘ (p)/(RT)) is derived. The total loss couples prediction, structure, docking and quantum Fisher regularization into a single objective L=L_"pred" +L_"struct" +L_"dock" +L_"QFIM", with L_"QFIM" proportional to tr(F(θ)^(-1)).

Candidate peptides are passed through a three-gate "physics + geometry + immunology" oracle. First, a quantum-geometric gate requires that the Fubini-Study distance between ∣ψ(x)⟩ and a centroid ∣ψ(P)⟩ of empirically validated immunogenic peptides satisfy d_"FS" (ψ(x),ψ(P))≤d^"\*" . Second, a thermodynamic gate requires that the effective free energy and dissociation constant meet minimum binding strength criteria, ΔG_"eff" ^∘ (x)≤ΔG^"\*" or equivalently K_d^"eff" (x)≤K_d^"\*" . Third, an immunogenicity gate requires that the calibrated probability exceed a threshold, I ̂(x)≥I^"\*" . Let the total number of candidates be N, with M peptides passing all three filters. In abstract quantum terms, a uniform superposition over all candidates is ∣Ψ_0⟩=1/√N ∑_(j=1)^N▒〖∣j⟩,which can be decomposed into "marked" and "unmarked" subspaces as ∣Ψ_0⟩=sin⁡θ" "∣Ψ_"good" ⟩+cos⁡θ" "∣Ψ_"bad" ⟩, where 〖sin⁡〗^2 θ=M/N. A Grover-like amplitude amplification operator G is defined as the product of an oracle O that flips the phase of marked states and a diffusion operator D that reflects about ∣Ψ_0⟩. After r iterations, the state becomes ∣Ψ_r⟩=G^r∣Ψ_0⟩=sin⁡((2r+1)θ)∣Ψ_"good" ⟩+cos⁡((2r+1)θ)∣Ψ_"bad" ⟩, and the probability of measuring a marked index is P_r=〖sin⁡〗^2 ((2r+1)θ).

When θ is small (few good candidates), the optimal number of iterations that maximizes P_r is approximately r_"opt" ≈π/4 √(N/M), but in the NISQ regime and in the presence of uncertainty in M, COLONYVAQ uses a small number of iterations (typically one to three) to reliably amplify the weight of marked peptides without over-rotation. In practice, this Grover-style step is simulated or approximated in a manner compatible with available hardware and serves to focus GMP peptide synthesis on a compact, high-confidence subset.

Within the set of marked peptides, residual ties are broken using a composite score S(x)=αK_q (x,P)+β" " σ" ⁣" ((I ̂(x)-I^"\*" )/τ_I )+γ" " σ" ⁣" ((K_d^"\*" -K_d^"eff" (x))/τ_K ), where K_q (x,P)=〖∣⟨ψ(x)∣ψ(P)⟩∣〗^2, τ_I and τ_K set the steepness of transitions, and σ is the logistic function. This expression makes explicit how similarity to known positive controls, modeled immune potency, and predicted binding strength jointly determine the final ranking used to define the COLONYVAQ-CRC peptide cargo for each patient.

Rationale for Combination with mFOLFOX6 or CAPOX and Nivolumab

Oxaliplatin and fluoropyrimidines are standard components of adjuvant therapy in stage III colorectal cancer and can induce immunogenic cell death, increasing the release of tumor antigens and danger signals, which in turn enhances dendritic cell activation and antigen cross-presentation. Nivolumab 3 mg/kg every 2 weeks blocks PD-1, preventing exhaustion and functional suppression of vaccine-induced and chemotherapy-released tumor-specific T cells. The quantum-classical COLONYVAQ-CRC engine is intended to maximize the quality of neoantigen targets; immunogenic chemotherapy increases antigen availability; and PD-1 blockade sustains T-cell effector function. The early phase I trial will test the safety and feasibility of this three-component strategy in the adjuvant MRD setting and generate preliminary immune and molecular response data.

ELIGIBILITY:
* Eligibility
* Inclusion Criteria

  * **Diagnosis / Histology**
  * Histologically confirmed adenocarcinoma of the colon or rectum.
  * Pathology report available for central or sponsor review (if requested), including:
  * Primary tumor site (colon vs rectum)
  * Grade of differentiation
  * Resection margins
  * **Stage and Surgical Status**
  * Pathologic stage III disease (any T, N1-2, M0) per AJCC 8th edition.
  * R0 resection of the primary tumor documented by operative and pathology reports (no macroscopic or microscopic residual tumor at margins).
  * No evidence of distant metastatic disease (M1) on staging imaging (CT chest/abdomen/pelvis ± MRI/PET per institutional standard) within a protocol-defined window (e.g., ≤8 weeks prior to enrollment).
  * Enrollment and treatment initiation planned within a protocol-defined timeframe after surgery (e.g., 4-12 weeks post-resection), allowing appropriate recovery.
  * **Molecular Subtype (MSS/pMMR)**
  * Tumor confirmed MSS or pMMR by local testing using one or more of the following:
  * IHC for MLH1, MSH2, MSH6, and PMS2
  * PCR-based MSI panel
  * NGS-based MSI/MMR assessment
  * No evidence of dMMR/MSI-H status or POLE ultramutated phenotype.
  * **High-Risk Recurrence Profile**
  * At least one protocol-defined high-risk feature, including one or more of the following:
  * Pathologic T4 tumor
  * Pathologic N2 nodal status (≥4 positive lymph nodes)
  * Positive postoperative ctDNA (MRD) by a validated tumor-informed assay within a protocol-defined window after surgery/chemotherapy initiation
  * Other protocol-specified high-risk features (e.g., lymphovascular invasion, perineural invasion, poorly differentiated histology, inadequate lymph node sampling), as defined in the protocol/statistical analysis plan
  * **Suitability for Standard Adjuvant Chemotherapy**
  * Candidate for oxaliplatin-based adjuvant chemotherapy with one of the following:
  * mFOLFOX6 every 14 days for ~6 months, **or**
  * CAPOX (XELOX) every 21 days for ~3-6 months
  * Chemotherapy regimen (mFOLFOX6 vs CAPOX) determined before enrollment and recorded as a stratification factor.
  * No contraindications to oxaliplatin, 5-fluorouracil, leucovorin, or capecitabine (e.g., severe DPD deficiency; prior severe 5-FU/capecitabine toxicity).
  * **Suitability for Nivolumab**
  * Eligible in the investigator's judgment to receive anti-PD-1 therapy (nivolumab 3 mg/kg IV every 2 weeks), including:
  * No history of severe (Grade ≥3) immune-related adverse events from prior immunotherapy
  * No active autoimmune disease requiring systemic immunosuppression
  * **Performance Status**
  * ECOG performance status 0-1 at screening.
  * **Adequate Organ and Marrow Function** (documented within 14 days prior to enrollment; no transfusions/growth factors solely to meet eligibility)
  * **Hematologic**
  * ANC ≥ 1.5 × 10⁹/L
  * Platelets ≥ 100 × 10⁹/L
  * Hemoglobin ≥ 9.0 g/dL (transfusions allowed if clinically indicated, but not solely to qualify)
  * **Hepatic**
  * Total bilirubin ≤ 1.5 × ULN (≤3 × ULN allowed for known Gilbert's syndrome if direct bilirubin is normal)
  * AST and ALT ≤ 2.5 × ULN
  * Alkaline phosphatase ≤ 2.5 × ULN (higher thresholds may be allowed for non-malignant causes per protocol)
  * **Renal**
  * Serum creatinine ≤ 1.5 × ULN **or** creatinine clearance ≥ 50 mL/min (Cockcroft-Gault or institutional standard)
  * **Biospecimen Availability (COLONYVAQ)**
  * Adequate tumor tissue available from resected primary tumor (and/or metastases if applicable), including one of the following:
  * Fresh frozen tissue (preferred), **or**
  * FFPE block(s), **or**
  * ≥15 unstained slides (or equivalent) suitable for DNA/RNA extraction
  * Matched normal sample (peripheral blood) available for germline DNA sequencing.
  * Willingness to provide additional blood samples for ctDNA, immune monitoring, and exploratory assays per schedule.
  * Pre-existing WES/RNA-seq may be accepted if meeting COLONYVAQ requirements per protocol.
  * **Neoantigen Suitability**
  * At least one predicted high-quality tumor neoantigen identified by the COLONYVAQ pipeline meeting prespecified criteria, including:
  * Strong predicted binding to patient-specific HLA alleles (e.g., Kd in an established binder range)
  * Evidence of tumor RNA expression of the source gene/allele
  * Prioritization by multi-algorithm immunogenicity scoring and passage through COLONYVAQ quantum-geometric, thermodynamic, and immunogenicity gates
  * **OR**
  * Availability of pre-manufactured GMP-grade neoantigen peptides with demonstrated in vitro immunogenicity and acceptable safety profile.
  * **Life Expectancy**
  * Investigator-estimated life expectancy ≥ 3 years in the absence of CRC recurrence.
  * **Contraception and Pregnancy**
  * **Women of childbearing potential (WOCBP)**
  * Negative serum or urine pregnancy test within 7 days prior to randomization
  * Agreement to use highly effective contraception during treatment and for a protocol-defined period after last dose (e.g., 5 months after last nivolumab and 6 months after last chemotherapy, or per label/institutional guidance)
  * **Men with partners of childbearing potential**
  * Agreement to use effective contraception and avoid sperm donation during treatment and for the protocol-defined period after last dose
  * **Informed Consent and Compliance**
  * Able to understand and voluntarily sign written informed consent.
  * Willing and able to comply with all study procedures (visits, imaging, blood draws, follow-up).
* Exclusion Criteria

  * **Residual or Metastatic Disease at Baseline**
  * R2 resection or indeterminate margins not clearly R0.
  * Radiologic or histologic evidence of distant metastases (M1) at baseline staging (e.g., liver, lung, peritoneum).
  * Gross residual disease at the primary site.
  * **Mismatch Repair-Deficient / MSI-High / POLE-Ultramutated Disease**
  * Known dMMR/MSI-H CRC or POLE ultramutated tumors for which checkpoint inhibition is standard/preferred.
  * **Prior Anticancer Therapy (Beyond Allowed Neoadjuvant)**
  * Prior systemic therapy for metastatic CRC.
  * Neoadjuvant chemotherapy/chemoradiotherapy that:
  * Was not completed within protocol-defined windows, **or**
  * Led to unresolved Grade ≥2 non-hematologic toxicity (excluding alopecia or clinically insignificant neuropathy, per protocol)
  * Prior tumor vaccine targeting TAAs or neoantigens (peptide, DC, viral, RNA, or DNA).
  * Prior immune checkpoint inhibitor therapy (anti-PD-1, anti-PD-L1, anti-CTLA-4).
  * **Active or Uncontrolled Infections**
  * Systemic infection requiring IV or oral antimicrobials that would interfere with study treatment per investigator judgment.
  * Uncontrolled HIV (e.g., CD4 below protocol threshold or unsuppressed viral load).
  * Active hepatitis B with HBV DNA above predefined limit, or active hepatitis C with detectable HCV RNA not adequately treated.
  * Other clinically significant infections posing excessive risk with immunotherapy, vaccine, or chemotherapy.
  * **Autoimmune Disease / Immunosuppression**
  * Severe/uncontrolled autoimmune disease requiring systemic immunosuppression (e.g., high-dose corticosteroids, biologics), including (examples):
  * Systemic lupus erythematosus
  * Inflammatory bowel disease with recent flares
  * Rheumatoid arthritis requiring biologics
  * Multiple sclerosis
  * Myasthenia gravis
  * Exceptions may include (per protocol):
  * Stable autoimmune thyroiditis on replacement therapy
  * Vitiligo
  * Well-controlled type 1 diabetes
  * Chronic systemic corticosteroids >10 mg prednisone equivalent daily (or other immunosuppressants) within a protocol-defined window prior to first dose (unless physiologic/adrenal replacement).
  * **Transplant History**
  * Prior allogeneic hematopoietic stem cell transplantation.
  * Prior solid organ transplantation (e.g., kidney, liver, heart).
  * **Hypersensitivity / Drug Intolerance**
  * Severe hypersensitivity (e.g., anaphylaxis) to any of the following:
  * COLONYVAQ-CRC components (peptides/excipients)
  * Poly I:C or similar TLR agonists
  * Nivolumab or other anti-PD-1/PD-L1 agents
  * Oxaliplatin, 5-FU, leucovorin, or capecitabine (including severe DPD deficiency)
  * **Concurrent Malignancy**
  * Active second primary malignancy requiring systemic therapy or expected to require systemic therapy during the trial.
  * Exceptions:
  * Adequately treated basal cell or squamous cell skin carcinoma
  * Cervical carcinoma in situ
  * Other malignancies in complete remission not expected to relapse or require systemic therapy within 5 years, per investigator judgment
  * **Significant Comorbidities**
  * Clinically significant/unstable cardiovascular disease, including:
  * MI within 6 months
  * Unstable angina
  * Uncontrolled arrhythmias
  * CHF NYHA class III-IV
  * Uncontrolled hypertension despite medical therapy
  * Stroke or TIA within 6 months (if risk is increased per investigator judgment).
  * Severe COPD or interstitial lung disease with significant impairment, or prior pneumonitis requiring systemic steroids.
  * Any other serious uncontrolled condition (e.g., poorly controlled diabetes, severe cirrhosis, advanced renal failure) that may compromise safety or adherence.
  * **Pregnancy / Lactation**
  * Pregnant at screening (positive pregnancy test).
  * Breastfeeding (must discontinue lactation before first dose).
  * **Concurrent Investigational Agents / Confounding Therapies**
  * Participation in another interventional trial with systemic investigational agents (unless sponsor/IRB-approved and not confounding).
  * Live attenuated vaccine within a protocol-defined period (e.g., 30 days) prior to first dose of nivolumab or COLONYVAQ-CRC, or during study treatment.
  * **Other Conditions Affecting Compliance or Assessment**
  * Psychiatric illness, cognitive impairment, substance abuse, or social situation limiting adherence to study requirements.
  * Any condition that, in the investigator's opinion, makes the participant unsuitable or interferes with interpretation of safety, immunologic, or clinical outcomes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2030-12-02 (Estimated); Study Completion 2031-12-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent AEs/SAEs and Immune-Related AEs (CTCAE v5.0) With COLONYVAQ-CRC Plus Chemotherapy and Nivolumab | From first dose of any study treatment (chemotherapy, vaccine, or nivolumab) through 90 days after the last dose (total observation ~12 months per patient).
  Incidence, nature, and severity (CTCAE v5.0 grade) of treatment-emergent adverse events (AEs) and serious adverse events (SAEs), with specific assessment of vaccine-attributable toxicities and immune-related adverse events. A prespecified safety expansion benchmark will be evaluated: among the first 12 patients, <3 with vaccine-related toxicity >Grade 2 and no vaccine-related Grade 4 toxicity prior to expansion from 12 to 50 patients.

SECONDARY OUTCOMES:
Feasibility of COLONYVAQ-CRC Vaccine Manufacturing and Delivery | From enrollment through completion of the prime vaccination phase, typically within the first 8 weeks after the first vaccine dose.
  Proportion of enrolled patients in whom adequate tumor and blood material can be obtained, neoantigen discovery and COLONYVAQ-based peptide prioritization can be completed, GMP manufacturing succeeds, and at least a predefined minimum number of vaccine doses are administered without major logistical failure.
Proportion of Participants With ≥2-Fold Increase in Neoantigen-Specific T Cells From Baseline | Baseline (within 28 days before the first vaccine dose), during vaccination at approximately Weeks 4, 12 and 20 after first vaccination, at the end of the vaccination period (around 8 months after first vaccination), and at a 12-month follow-up.
  Change from baseline in COLONYVAQ-selected neoantigen peptide-specific CD4⁺ and CD8⁺ T-cell responses measured in peripheral blood. Responses will be assessed using IFN-γ ELISPOT, intracellular cytokine staining (ICS), and/or peptide-MHC multimer staining. The outcome is reported as the percentage of participants who demonstrate a ≥2-fold increase over baseline in neoantigen-specific T cells at any post-baseline time point.
ctDNA Clearance at End of Adjuvant Chemotherapy | Postoperative baseline before adjuvant therapy (within 4 weeks prior to the first chemotherapy cycle), during treatment at approximately 3 months and at the end of adjuvant chemotherapy, around 7 months after randomization, and at follow-up at 12 months.
  Description: Among participants with detectable postoperative baseline ctDNA, the proportion (%) who convert to undetectable ctDNA at the end of adjuvant chemotherapy.
  Measurement tool/parameter: Circulating tumor DNA status (detectable vs undetectable) measured by a validated ctDNA assay (tumor-informed or tumor-agnostic platform, as specified in the protocol).
Preliminary Disease-Free Survival (DFS) | From the date of first study treatment until first documented recurrence of colorectal cancer or death from any cause, whichever occurs first, with planned descriptive analysis at 36 months after first patient first treatment.
  DFS will be estimated using Kaplan-Meier methods in this single-arm cohort. Because this is a phase I study, DFS results are considered exploratory and will be used to inform assumptions and endpoint definitions for subsequent phase II trials rather than to draw definitive efficacy conclusions.
Preliminary Overall Survival (OS) | From the date of first study treatment until death from any cause, with follow-up planned up to 60 months after the first patient starts treatment.
  OS will be summarized descriptively with Kaplan-Meier estimates. As with DFS, OS data will be hypothesis-generating and used to shape the design of later-phase studies.
Health-Related Quality of Life (HRQoL) | Baseline within 28 days before first chemotherapy or first vaccine dose, at the end of adjuvant chemotherapy approximately 6 months after treatment initiation, at 12 months, and annually thereafter up to 36 months.
  Change from baseline in global health status and selected functional and symptom scales measured by EORTC QLQ-C30 (and, optionally, colorectal cancer-specific modules such as QLQ-CR29). Results will be compared over time within the cohort to assess the impact of the combination regimen on quality of life.
Breadth of Neoantigen-Specific T-Cell Responses (Number of Reactive Peptides per Participant) | Baseline (within 28 days before the first vaccine dose), during vaccination at approximately Weeks 4, 12 and 20 after first vaccination, at the end of the vaccination period (around 8 months after first vaccination), and at a 12-month follow-up.
  Breadth of COLONYVAQ-selected neoantigen peptide-specific CD4⁺ and CD8⁺ T-cell responses measured in peripheral blood using IFN-γ ELISPOT, ICS, and/or peptide-MHC multimer staining. The outcome is reported as the number of neoantigen peptides per participant that elicit a measurable T-cell response at post-baseline time points.
Persistence of Neoantigen-Specific T-Cell Responses Over Time | Baseline (within 28 days before the first vaccine dose), during vaccination at approximately Weeks 4, 12 and 20 after first vaccination, at the end of the vaccination period (around 8 months after first vaccination), and at a 12-month follow-up.
  Durability of COLONYVAQ-selected neoantigen peptide-specific CD4⁺ and CD8⁺ T-cell responses in peripheral blood assessed longitudinally by IFN-γ ELISPOT, ICS, and/or peptide-MHC multimer staining. The outcome is reported as the proportion of participants with a measurable neoantigen-specific T-cell response maintained at prespecified follow-up visits (e.g., sustained response at consecutive time points after first detection).
ctDNA Clearance at 12 Months | Postoperative baseline before adjuvant therapy (within 4 weeks prior to the first chemotherapy cycle), during treatment at approximately 3 months and at the end of adjuvant chemotherapy, around 7 months after randomization, and at follow-up at 12 months.
  Description: Among participants with detectable postoperative baseline ctDNA, the proportion (%) who have undetectable ctDNA at 12 months.
  Measurement tool/parameter: Circulating tumor DNA status (detectable vs undetectable) measured by the study ctDNA assay.
Density of Tumor Immune Cell Infiltrates | Baseline (within 28 days before the first vaccine dose), during vaccination at approximately Weeks 4, 12 and 20 after first vaccination, at the end of the vaccination period (around 8 months after first vaccination), and at a 12-month follow-up.
  Description: Quantification of intratumoral immune cell infiltrates (e.g., CD8⁺ T cells, regulatory T cells, macrophage subsets) in available tumor tissue.
  Measurement tool: Immunohistochemistry (IHC) and/or multiplex immunofluorescence (mIF).
  Unit of measure: Cell density (e.g., cells/mm²) and/or % of total nucleated cells, as defined by the assay readout.

OTHER OUTCOMES:
T-Cell Receptor (TCR) Clonotype Diversity, Expansion, and Persistence | Baseline within 28 days prior to first vaccine dose, during vaccination at Weeks 4, 12, and 20 after first vaccination, at the end of the vaccination period approximately at 7 months, and at 12 and 24 months after initiation of adjuvant therapy.
  Analysis of TCR clonotype repertoires from peripheral blood mononuclear cells (and optionally from tumor tissue when available), using bulk or single-cell TCR sequencing. Endpoints include diversity indices, expansion of clonotypes associated with COLONYVAQ targets, and persistence of these clonotypes over time. Correlations between TCR dynamics, quantum-classical selection scores (for example K_q, ΔG_"eff" ^∘, K_d^"eff" , I ̂(p)), and clinical outcomes will be explored.
Correlation of Tumor Immune Features With Vaccine-Induced Systemic Immune Responses | Baseline resection specimen (pre-treatment) and optional tissue samples at recurrence or predefined timepoints up to 60 months after treatment initiation.
  Description: Correlation between tumor immune features (Outcome Measures 1-3) and vaccine-induced systemic immune responses measured in peripheral blood.
  Measurement tools:
  Tumor immune features assessed by IHC/mIF (cell densities/percentages; PD-L1 scoring) and transcriptomic profiling (signature scores).
  Systemic immune responses assessed by prespecified immune assays (e.g., IFN-γ ELISPOT, intracellular cytokine staining, and/or peptide-MHC multimer staining).
  Unit of measure: Correlation coefficient (e.g., Spearman's ρ or Pearson's r, prespecified).
Clinical Correlation of Genomic and COLONYVAQ Modeling Features With Immune Response Breadth and Clinical Outcomes | Baseline molecular profiling performed before vaccine manufacture, with clinical and immune outcomes followed up to 60 months after treatment initiation.
  Clinical endpoints used in correlative analyses include:
  ctDNA response measured by the study ctDNA assay (e.g., clearance or quantitative change, per protocol definition) (unit: % with clearance and/or quantitative ctDNA change in assay units).
  Disease-free survival (DFS) (unit: time-to-event, e.g., months). Overall survival (OS) (unit: time-to-event, e.g., months).
Quantum-Geometric Descriptor Values From the COLONYVAQ Quantum Model | From baseline vaccine design (pre-treatment) through longitudinal immune monitoring at approximately Weeks 4, 12, 20, 7-8 months, and at 12 and 24 months after first vaccine dose.
  Description: Retrospective quantification of quantum-geometric descriptors generated by the COLONYVAQ quantum modeling framework, including Fubini-Study distance (d_FS), quantum kernel value K_q(x,y), entanglement entropy, and quantum Fisher information (QFI)-based regularization terms.
  Measurement tool: COLONYVAQ quantum modeling pipeline / computational feature extraction.
  Unit of measure: Descriptor values in model-defined units (e.g., d_FS distance units; K_q(x,y) kernel value; entropy units; QFI-based term value), as output by the model.
Vaccine-Induced Neoantigen-Specific T-Cell Immunogenicity | From baseline vaccine design (pre-treatment) through longitudinal immune monitoring at approximately Weeks 4, 12, 20, 7-8 months, and at 12 and 24 months after first vaccine dose.
  Description: Vaccine-induced neoantigen-specific T-cell responses in peripheral blood.
  Measurement tool: Prespecified immunogenicity assays (e.g., IFN-γ ELISPOT, intracellular cytokine staining, and/or peptide-MHC multimer staining).
  Unit of measure: Immune response magnitude and/or frequency in assay-specific units (e.g., spot-forming units, % cytokine-positive T cells, % multimer-positive T cells), as defined in the protocol.
ctDNA Molecular Response (Detectable vs Undetectable) for Retrospective Modeling | From baseline vaccine design (pre-treatment) through follow-up at ~Weeks 4, 12, 20, ~7-8 months, and 12 and 24 months after first vaccine dose.
  Description: Proportion of participants with ctDNA response, defined as conversion from detectable ctDNA at baseline to undetectable ctDNA at a post-baseline timepoint, assessed by the study ctDNA assay.
  Unit of Measure: Percentage (%) of participants with ctDNA response.
Change in ctDNA Quantitative Level for Retrospective Modeling | From baseline vaccine design (pre-treatment) through follow-up at ~Weeks 4, 12, 20, ~7-8 months, and 12 and 24 months after first vaccine dose.
  Description: Change from baseline in quantitative ctDNA level measured by the study ctDNA assay (e.g., ctDNA fraction/VAF or ctDNA concentration, per assay output), evaluated at each timepoint for retrospective model performance analyses.
  Unit of Measure: Assay-specific quantitative units (e.g., VAF [%] or copies/mL), as reported by the ctDNA assay.
Disease-Free Survival (DFS) for Retrospective Modeling | From first vaccine dose through 24 months after first vaccine dose.
  Description: DFS defined as time from first vaccine dose to first documented disease recurrence/progression or death from any cause, per protocol definition, used in retrospective model performance analyses.
  Unit of Measure: Time-to-event (months).
Overall Survival (OS) for Retrospective Modeling | From first vaccine dose through 24 months after first vaccine dose.
  Description: OS defined as time from first vaccine dose to death from any cause, per protocol definition, used in retrospective model performance analyses.
  Unit of Measure: Time-to-event (months).

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Grigoriadis, Pharmacist PharmD, Principal Investigator — Biogenea Pharmaceuticals Ltd.
Locations (1):
- Biogenea Pharmaeuticals Ltd, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the COLONYVAQ-CRC platform and its underlying quantum-classical neoantigen selection methods are the subject of an ongoing patent application. Data sharing will be reconsidered after the patent process is complete and the associated intellectual property protections are clarified.